CLINICAL TRIAL: NCT04300283
Title: A Pilot Study Investigating the Feasibility of a Pre-operative Hypnosis Intervention to Prevent Post-operative Pain After Thoracic and Breast Cancer Surgery
Brief Title: Pre-operative Hypnosis to Prevent Side Effects After Surgery
Acronym: PREVENTpilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Silje Endresen Reme, Professor, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2018/781
Record Dates: First submitted 2020-01-29; First posted 2020-03-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Breast Cancer Surgery
MeSH Terms: interventions — Hypnosis

STUDY DESIGN:
Intervention Model Description: Pilot testing of a pre-operative hypnosis intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pre-operative hypnosis (Experimental)
  Interventions: Behavioral: Hypnosis

INTERVENTIONS:
Behavioral: Hypnosis — See previous description

SUMMARY:
The aim of the pilot study is to translate and feasibility test a brief hypnosis intervention in 8-10 patients that are about to undergo thoracic surgery and in 4-5 patients about to undergo breast cancer surgery.

DETAILED DESCRIPTION:
The hypnosis intervention will be based on a protocol from Montgomery et al. They showed in a recent study that a brief 15-minute hypnosis intervention was effective in reducing a number of common side effects, including pain, fatigue and nausea. The scripted session includes a relaxation-based induction, suggestions for pleasant visual imagery, suggestions to experience relaxation and peace, and specific symptom-focused suggestions. The intervention will be professionally translated into Norwegian, and adapted and modified as necessary to the specific context of this study. The PI, who is a an experienced clinical psychologist, will hold the session in the pilot study. Patients will further be instructed to use hypnosis on their own following the intervention session.

The patients will further be invited to participate in semi-structured interviews upon completion of the intervention, either by phone or in person, to discuss their experiences with the intervention, and share any advice for modifications or changes to the interventions or procedures. Systematic text condensation will be applied in the analyses of the interviews.

ELIGIBILITY:
Inclusion Criteria:

* Patients about to undergo either breast cancer surgery or thoracic surgery

Exclusion Criteria:

* Insufficient Norwegian speaking or writing skills to participate in the intervention
* cognitive and psychiatric impairment
* other serious malignancies

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Patient experiences of the intervention | 1 week post-surgery
  Obtained through qualitative interviews to assess patient experiences and possibly adverse effects of the intervention

SECONDARY OUTCOMES:
NRS Pain intensity one week after surgery | 1 week post-surgery
  Numeric Rating Scale (0-10) of pain intensity in the surgical and referred area
Fatigue severity one week after surgery | 1 week post-surgery
  Numeric Rating Scale of fatigue severity

CONTACTS AND LOCATIONS:
Overall Officials: Silje E Reme, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lind SB, Jacobsen HB, Solbakken OA, Reme SE. Clinical Hypnosis in Medical Care: A Mixed-Method Feasibility Study. Integr Cancer Ther. 2021 Jan-Dec;20:15347354211058678. doi: 10.1177/15347354211058678. PMID 34818921